CLINICAL TRIAL: NCT02550145
Title: The Role of GLP-1 in Mediating Glucose Reductions After Bariatric Surgery
Brief Title: Role of GLP-1 in Hyperinsulinemic Hypoglycemia Post-bariatric Surgery
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Tracey McLaughlin (Other)
Responsible Party: Sponsor-Investigator, Tracey McLaughlin, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 29010
Record Dates: First submitted 2015-06-05; First posted 2015-09-15 (Estimated); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Hypoglycemia
Keywords: Hyperinsulinemic; post-bariatric surgery
MeSH Terms: conditions — Hypoglycemia | interventions — exendin (9-39)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exendin(9-39) (Experimental): IV infusion of Exendin (9-39).
  Interventions: Drug: Exendin (9-39)
- Placebo (Placebo Comparator): IV infusion of normal saline
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Exendin (9-39) — IV infusion of Exendin (9-39) during standardized oral glucose tolerance test (OGTT).
  Arms: Exendin(9-39)
Other: Placebo — IV infusion of Placebo (normal saline) during standardized oral glucose tolerance test (OGTT)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the role of GLP-1 in causing extreme postprandial glucose reductions after bariatric surgery in a subset of patients who have severe symptomatic hypoglycemia.

DETAILED DESCRIPTION:
The physiologic mechanisms mediating the glucose-lowering effect of Roux-en-Y Gastric Bypass (RYGB) or post-Vertical Sleeve Gastrectomy (VSG) are unknown. The reduction in glucose excursions prior to weight loss has lead to postulates that the incretin hormone, GLP-1, may play an important role.

The purpose of this study is to evaluate the role of GLP-1 in causing extreme postprandial glucose reductions in a subset of post-bariatric patients through the pharmacologic blockade of the GLP-1 receptor in post-RYGB or post-VSG patients with severe symptomatic hypoglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18-65
* BMI 25-40 with a clinical diagnosis of severe symptomatic hypoglycemia after bariatric surgery

Exclusion Criteria:

* Acute medical illness, such as acute bacterial or viral syndrome, febrile illness, acute abdominal symptoms, orthopedic injury within one week
* History of cardiac failure, renal insufficiency (estimated Crcl<30cc/min), hepatic insufficiency, chronic obstructive pulmonary disease, anemia (Hct<30%), or uncontrolled hypertension (SBP>160 or DBP>100)
* Pregnancy
* Use of medications that affect glucose metabolism
* Fasting glucose >150 or HbA1c>7.5 on Metformin
* Women of childbearing potential (will have a pregnancy test, in addition use of abstinence for at least one month prior to study or use two types of contraceptives, hormonal implant or Depo Provera)
* Active, uncontrolled psychiatric disease
* Participating in other studies or have received investigational medications within the past month or 5 half-lives of the drug, whichever is longer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Plasma glucose area under the curve | 0 to 180 minutes

SECONDARY OUTCOMES:
Plasma insulin area under the curve | 0 to 180 minutes

OTHER OUTCOMES:
Hypoglycemia symptom score | 0-180 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Craig, M.D., Study Director — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Craig CM, Liu LF, Deacon CF, Holst JJ, McLaughlin TL. Critical role for GLP-1 in symptomatic post-bariatric hypoglycaemia. Diabetologia. 2017 Mar;60(3):531-540. doi: 10.1007/s00125-016-4179-x. Epub 2016 Dec 14. PMID 27975209